CLINICAL TRIAL: NCT02501018
Title: A Prospective, Open Label, Controlled, Randomized, Multicenter Study to Assess the Efficacy and Safety of CLBS12 in Patients with Critical Limb Ischemia (CLI) Due to Arteriosclerosis Obliterans (ASO) with a Single-arm Substudy to Assess the Safety and Potential Efficacy of CLBS12 in Patients with CLI Due to Buerger's Disease (BD)
Brief Title: Study to Assess the Efficacy and Safety of CLBS12 in Patients with Critical Limb Ischemia (CLI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLBS12-P01
Record Dates: First submitted 2015-07-14; First posted 2015-07-17 (Estimated); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Critical Limb Ischemia; Buerger Disease; Thromboangiitis Obliterans; Atherosclerosis Obliterans
Keywords: CLI, ASO, TAO
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Thromboangiitis Obliterans | interventions — betibeglogene autotemcel; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CLI Due to ASO with CLBS12 + SOC (Experimental): This group of subjects with CLI due to ASO will be administered with CLBS12 + SOC for collecting efficacy and safety data.
  Interventions: Biological: CLBS12; Drug: SOC
- CLI Due to ASO with SOC (Active Comparator): This group of subjects with CLI due to ASO will be administered with SOC only.
  Interventions: Drug: SOC
- CLI Due to BD with CLBS12 (Experimental): CLBS12 will be administered to patients with CLI due to BD for collecting safety and efficacy data.
  Interventions: Biological: CLBS12; Drug: SOC

INTERVENTIONS:
Biological: CLBS12 — Intramuscular transfusion of CLBS12.
  Other Names: CD34+ cells
  Arms: CLI Due to ASO with CLBS12 + SOC; CLI Due to BD with CLBS12
Drug: SOC — Standard of care (SOC) is defined as pharmacotherapy with approved drugs (e.g., antiplatelets, anticoagulants, and vasodilators including prostanoids).
  Other Names: Standard of care

SUMMARY:
A prospective, open label, controlled, randomized, double arm, multi-center study to assess the efficacy and safety of CLBS12 in patients with critical limb ischemia (CLI) due to arteriosclerosis obliterans (ASO) with a single arm sub-study to assess the safety and potential efficacy of CLBS12 in patients with CLI due to Buerger's Disease (BD).

DETAILED DESCRIPTION:
Main ASO Study: This study will compare safety and efficacy of intramuscular transplantation of autologous CD34+ cells (CLBS12) plus standard of care (SOC) pharmacotherapy (cell treatment arm) versus SOC pharmacotherapy alone (e.g., antiplatelets, anticoagulants, and vasodilators including prostanoids) (control arm) in subjects with CLI categorized as Rutherford score 4 or 5 due to ASO aged 20 to 85 years and with no endovascular or surgical revascularization options. Subjects assigned to the cell treatment arm will continue SOC pharmacotherapy and will also receive subcutaneous injections of GRAN® 5 ug/kg/day for 5 days and undergo apheresis on the last day of GRAN® administration. Then each subject in the cell treatment arm will receive intramuscular injections of autologous CD34+ cells. Subjects assigned to the control arm will continue to receive SOC pharmacotherapy alone with the possibility of receiving cell treatment via the rescue option.

BD Substudy: A single arm substudy is included to assess the safety and efficacy of intramuscular transplantation of CLBS12 in patients (N=~5) with CLI categorized as 4 or 5 Rutherford score due to BD aged 20 to 85 years. Subjects who give informed consent will be screened for eligibility within 28 days before registration. Subjects will continue SOC pharmacotherapy and will also receive subcutaneous injections of GRAN® 5 µg/kg/day for 5 days (Pretreatment Days 1 5) to mobilize CD34+ cells into the peripheral blood and undergo apheresis on pretreatment Day 5 to collect CD34+ cells. The choice of pharmacotherapy will be made by the investigators.

Each subject in a cell treatment arm will receive intramuscular injections of up to 1 × 10^6 autologous CD34+ cells/kg/limb. All subjects will be evaluated for efficacy and safety assessments during approximately 12 months.

Efficacy assessments include CLI free status, AFS, PFS, ABI, TBI, SPP, TcPO2, ICD, VAS, and AQA.

ELIGIBILITY:
Inclusion Criteria:

* subject has CLI caused by ASO or BD

Exclusion Criteria:

* < 20 years old

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Time to continuous CLI-free status | 1 year
  CLI-free is determined by assessing the Rutherford score (</=3) by the investigator and a central adjudication committee.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen K Buck, MD, Study Director — Lisata Therapeutics, Inc.
Locations (12):
- Japan (12):
  - Asahikawa Medical University Hospital - 1-1-1 Higashi-2jou, Midorigaoka, Asahikawa-shi
  - Fukuoka Sanno Hospital, Fukuoka
  - Shonan Kamakura General Hospital, Kamakura
  - Kobe City Medical Center General Hospital, Kobe
  - Shinsuma General Hospital, Kobe
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - Oita Oka Hospital, Ōita
  - Nippon Medical School Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Toho University Medical Center Ohashi Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Women's Medical University, Tokyo

IPD SHARING:
Plan to Share IPD: No